CLINICAL TRIAL: NCT00760734
Title: HBOT in Chronic Traumatic Brain Injury/Post Concussion Syndrome and TBI/PTSD Pilot Trial
Brief Title: Hyperbaric Oxygen Therapy (HBOT) in Chronic Traumatic Brain Injury (TBI)/Post Concussion Syndrome (PCS) and TBI/Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paul G. Harch, M.D. (Other)
Collaborators: Semper Fi Fund (Unknown); Marine Corps-Law Enforcement Foundation (Other); Coalition to Support America's Heroes (Unknown); Thirty-eight other contributors (Unknown)
Responsible Party: Sponsor-Investigator, Paul G. Harch, M.D., Clinical Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSU IRB #7051
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: TBI (Traumatic Brain Injury); Post Concussion Syndrome; Post Traumatic Stress Disorder; Chronic Post Traumatic Stress Disorder
Keywords: Chronic traumatic brain injury; Post concussion syndrome; Post traumatic stress disorder; Chronic post traumatic stress disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperbaric oxygen therapy-TBI/PCS (Experimental): Intervention: Low pressure hyperbaric oxygen therapy, 40 or 80 twice daily, 5d/week, HBOTs at 1.5 ATA/60 minutes each. One month no treatment period between the 40th and 41st HBOT
  Interventions: Drug: Low pressure hyperbaric oxygen therapy
- Hyperbaric Oxygen Therapy-PCS/PTSD (Experimental): Intervention: Low pressure hyperbaric oxygen therapy, 40 or 80 twice daily, 5d/week, HBOTs at 1.5 ATA/60 minutes each. One month no treatment period between the 40th and 41st HBOT
  Interventions: Drug: Low pressure hyperbaric oxygen therapy

INTERVENTIONS:
Drug: Low pressure hyperbaric oxygen therapy — HBOT at 1.5 ATA/60 minutes twice/day, five days/week for 40 or 80 treatments
  Other Names: HBOT
Drug: Low pressure hyperbaric oxygen therapy — HBOT: 1.5 ATA/60 minutes twice/day, 5 days/week for 40 or 80 treatments
  Other Names: HBOT

SUMMARY:
This is a pilot trial to see if one or two 40 treatment courses of low pressure hyperbaric oxygen therapy can improve cognition and brain imaging in subjects with either chronic mild-moderate traumatic brain injury (TBI), also known as post-concussion syndrome (PCS) or chronic PCS with post-traumatic stress disorder (PTSD) secondary to blast injury.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-65 years old
* One or more mild-moderate TBI's characterized by loss of consciousness due to blast injury that is a minimum of one year old and occurred after 9/11/2001
* Absence of acute cardiac arrest or hemorrhagic shock at time of TBI.
* Absence of intracranial neurosurgery post-TBI
* Disability Rating Scale of 0-3
* Negative Michigan Alcohol Screening Test (MAST)
* Negative Drug Abuse Screening Test (DAST)
* Negative urine toxicology screen for drugs of abuse
* Negative pregnancy test in females
* Otherwise good health
* Less than 90% on the Percent Back to Normal Rating Scale

Exclusion Criteria:

* Pulmonary disease that precludes HBOT
* Unstable medical conditions that are contraindicated in HBOT
* Severe confinement anxiety
* Pregnancy
* Other pre-TBI neurological diagnoses
* Pre or post TBI history of substance abuse
* Pre or post TBI history of alcoholism.
* Participation in another experimental trial with active intervention.
* High probability of inability to complete the experimental protocol.
* Previous HBOT
* History of hospitalization for past TBI, stroke, nonfebrile seizures, or any seizure history other than seizure at the time of TBI
* Past or current history of mental retardation (baseline FSIQ < 71.
* Pre/post-TBI history of systemic illness with impact on CNS (P.I.'s decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Psychometric testing | 30 days

SECONDARY OUTCOMES:
SPECT brain imaging | 30 days
Quality of life measurements | 30 days
Return to school or work | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Harch, M.D., Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- LSU Health Sciences Center, New Orleans, Louisiana, United States

REFERENCES:
- [Result] Harch PG, Andrews SR, Fogarty EF, Amen D, Pezzullo JC, Lucarini J, Aubrey C, Taylor DV, Staab PK, Van Meter KW. A phase I study of low-pressure hyperbaric oxygen therapy for blast-induced post-concussion syndrome and post-traumatic stress disorder. J Neurotrauma. 2012 Jan 1;29(1):168-85. doi: 10.1089/neu.2011.1895. Epub 2011 Nov 22. PMID 22026588